CLINICAL TRIAL: NCT02488343
Title: Personal Profile of Adherence to Therapy and Tailored Interventions to Promote Adherence in Multiple Sclerosis Patients
Brief Title: Profile of Adherence to Therapy and Interventions to Promote Adherence in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ariel Miller, Director of Multiple Sclerosis & Brain Research Center, Carmel Medical Center, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMC-14-0061-CTIL
Record Dates: First submitted 2015-06-28; First posted 2015-07-02 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Adherence; Therapies; Psychological Intervention
MeSH Terms: conditions — Multiple Sclerosis | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Intervention (Experimental): Participants in this group will receive tailored psychological intervention to promote adherence to their drug therapy.
  Interventions: Behavioral: Behavioral Intervention
- Non Intervention group (No Intervention): Participants in this group will be observed but will not receive any intervention.

INTERVENTIONS:
Behavioral: Behavioral Intervention — Three types of intervention will be used: a) Interventions aimed to dealing with cognitions and habits will be based on cognitive-behavioral therapy (CBT) principles. b) Interventions aimed to dealing with affective factors that interfere with adherence will be based on dynamic therapy, crisis intervention and supportive elements. c) In the case of condition-related or therapy related barriers to adherence, psycho-educational multidisciplinary interventions of 1-2 appointments will be offered. Education about injection techniques and about reasonable expectations from therapy, and from MS itself, are a key strategy to successfully maintaining adherence.
  Arms: Behavioral Intervention

SUMMARY:
Adherence is an active process wherein the patient acts in collaboration with the medical and paramedical staff in order to improve his/her health. Adherence to medication comprises of implementation and persistence and it is estimated to be around 50% in various chronic illnesses, including Multiple Sclerosis (MS). MS patients who fail to properly adhere to their DMTs regimen may be at increased risk for the development of new central nervous system lesions, exacerbations, increased disabilities and poorer quality of life. Plausible reasons for the low adherence rates in MS mentioned in the literature include patients' attributes, condition attributes and therapy related factors.

The objective of this study is to develop a personal profile of adherence based in the factors mentioned above. In the first part of the study patients will be followed up and the profile My Multiple Sclerosis Perception Adherence Scoring System (MyMS_PASS) will be created and tested. In the second part, patients with non-optimal rates of adherence will receive tailored intervention in order to improve therapy to treatment. This work may serve as a model for the study of adherence to therapy and the development of interventions in MS as well as in other chronic diseases.

DETAILED DESCRIPTION:
Background Adherence is an active process wherein the patient acts in collaboration with the medical and paramedical staff in order to improve his/her health. Adherence to medication comprises of implementation and persistence and it is estimated to be around 50% in various chronic illnesses. Lack of persistence is the greater impediment to adherence in most cases (drops to approximately 60% over the course of a year). Non-adherence to prescribed treatment increases the frustration of both the patient and provider and can increase health care costs, including unnecessary hospitalizations and illness exacerbation.

A review of the World Health Organization (WHO) on adherence to therapy reveals a dynamic and complex issue associated simultaneously with several factors: social and economic factors, factors related to the health care team/system, characteristics of the disease, characteristics of the disease therapies and patient-related factors. In this latter category of patient-related issues this review identifies the following as major barriers: lack of information and skills, low motivation and self-efficacy, and lack of support for behavioral changes. Other patient related issues that influence adherence include patients' attributes: affective attributes (depression and anxiety) and cognitive attributes (illness- relevant cognition, perceptions of disease factors, and beliefs about treatment). The review emphasizes that low adherence is not a given fact and because of its vast significance, the WHO targeted it as "the best investment for tackling chronic conditions effectively" . Phillips, Leventhal & Leventhal propose to add two processes that occur after behavior initiation that are theorized to contribute to prediction of long term medication adherence: 'coherence' of patients' beliefs from experiences with treatment and habit development.

Multiple Sclerosis (MS) is the most common neurologic disease affecting young adults and can lead to severe physical disability and handicap.

Research on adherence in MS indicates adherence rates similar to those of other chronic illnesses, namely hovering around 50% two years after beginning of treatment. Patients who fail to properly adhere to their Disease Modifying Therapies (DMTs) regimen may be at increased risk for the development of new central nervous system lesions, exacerbation, and poorer quality of life.

Plausible reasons for the low adherence rates in MS mentioned in the literature include patients' attributes, condition attributes and therapy related factors:

Among patients' attributes, the research indicates 2 affective attributes that can be related to low adherence in MS: high prevalence of depression and anxiety. Research on cognitive attributes indicates an association between illness' perception, perceptions of medication and adherence in general, but to our knowledge, there's no research directly addressing this issue. To our knowledge, there's no research on habit strength and adherence, although habit strength was found predictive of low adherence in asthma patients and in patients with hypertension.

Among the condition-related factors that should be considered in MS adherence are the relapsing-remitting nature of the disease (medicines sometimes prescribed when the patient feels well). There is evidence that patients with few observable symptoms are typically less likely to adhere to complex medication regimens. Hancock and co-researchers found that patients with relatively stable disease were more likely to demonstrate poor medication adherence and poor appointment adherence.

Among the therapy related factors, 32% of non-adherence can be explained by the injection mode of delivery. Until recently the only available DMTs in MS included three preparations of beta interferon and glatiramer acetate. These therapies are all injected on a regular basis and associated with immediate undesirable results: painful site reactions, flu-like symptoms, increased spasticity, depression, and fatigue in a significant percentage of patients. In addition, the non-direct effect of the agents (unlike painkillers) might be one of the explanations for poor adherence. Recently, the FDA approved new DMTs for MS that are taken orally. Although it is plausible that adherence rates would improve with medications taken orally as opposed to injected medicines, there is some evidence to the contrary: for instance, Mohr and co-researchers found that soreness at injection site was related to continuing therapy; and Cramer found that patients with diabetes tend to be more adherent to injected therapy than to oral drugs. Thus, adherence factors may be different in injected and oral therapy, and it is important to study adherence in these two modalities.

We propose adherence to medication as a mediating variable between adjustment to MS and health outcomes. To our knowledge, there is no research addressing directly the issue of psychological interventions to promote adherence in MS. Significance This study will examine factors known in the literature as affecting adherence to therapy in MS or in other chronic illnesses in order to create a personal profile of adherence. This profile will allow the development of interventions tailored to the personal needs and barriers of patients regarding adherence. Improved adherence is expected to ensure treatment efficacy and may prevent irreversible tissue damage, resulting in prevention of accumulating functional disability. This work may serve as a model for the study of adherence to therapy and the development of interventions in other chronic diseases.

Design 400 patients treated with or planned to begin treatment with injected or oral therapy approved by the Israeli Ministry of Health for the treatment of MS will be recruited in "Carmel" MS Center.

The proposed study will consist of 4 phases:

1. Personal profile - In order to better understand therapy adherence in patients with MS, a personal profile of patient's attributes, condition and history of therapy, which takes into account the factors related to adherence mentioned above, will be gathered through questionnaires. This profile will be called MyMS_PASS (My Multiple Sclerosis Perception Adherence Scoring System).
2. Implementation and persistence -This phase includes tracking for 9 to 12 months the patients' personal profiles, habits and coherence between expectations and reality.
3. Intervention - According to the profiles assigned in phase 1 and the rates of adherence to therapy assessed in phase 2, all patients with the lowest adherence rates to therapy will be offered an intervention in the modality of Motivational Interviewing (MI) with a small psycho-educational component. The intervention will be tailored to the person's factors found as barriers to adherence. All non-adherent patients will be enrolled in an intervention, and their adherence - pre and post intervention - will be compared. The intervention will be applied by a health psychologist. The content of 5-10% of the meetings will be recorded in order to afford fidelity analysis (i.e., that the intervention delivered was as intended).
4. Evaluation of the intervention- Interventions will be evaluated by determining adherence to therapy and other relevant variables at baseline and at the end of the study for all participants in the study. Adherence to therapy before and after the intervention in the study and the control groups will be compared.

Study visits for data collection: Visit 1: Baseline- evaluation of illness and medication perception, adherence and habits.

Visit 2: About 6 months after beginning of follow-up- evaluation of illness and medication perception, adherence, habits and experiences with psychological interventions Visit 3: About 9 to 12 months after beginning of follow-up- Evaluation of adherence to therapy and of the factors related to adherence. By the end of this period intervention will be offered to patients that exhibit low adherence rates.

Visit 4: About 12 months after initiation of the intervention. Evaluation of adherence, habits, depression and anxiety and quality of life, for all participants in the study.

Proposed questionnaires:

1. Personal Information Questionnaire
2. Brief Illness Perception Questionnaire (BIPQ)
3. Beliefs about Medicines Questionnaire (BMQ)
4. Multiple Sclerosis Treatment Experience Questionnaire (MS-TEQ)
5. The Self-Report Habit Index (SRHI)
6. Questions about psychological intervention
7. Adult Dispositional Hope Scale (ADHS)
8. Hospital Anxiety and Depression Scale (HADS)
9. The World Health Organization Quality Of Life (WHOQOL-BREF)
10. Clinical questionnaire (EDSS) (for clinician)
11. Clinical follow-up questionnaire (EDSS) (for clinician)
12. Probabilistic Medication Adherence Scale (ProMAS)

Study Population MS patients visiting the MS center clinic at the Carmel Medical Center, treated or planned to begin treatment with injected or oral DMT for MS.

. Patients Recruitment MS patients visiting the MS center clinic at the Carmel Medical Center and responding to the inclusion criteria will be invited to participate in this study. Participants will receive an explanation from Prof. Miller, or the attending neurologist authorized by Prof Miller to do so, on the study aims and protocol. Patients who agree to participate will sign an informed consent. Information regarding their personal and family medical history, including data such as education and occupation, demographic and ethnicity data will be collected via questionnaires. In addition, several questionnaires related to adherence to treatment and patient's perception of treatment, disease and health will also be filled by the participants during the study visits, as described in the table "Proposed questionnaires" above. Medical staff will fill clinical questionnaires detailing patient clinical status including adverse events at each study visit. Data will also be collected from medical records, as necessary. Data collected through participants and physician filled forms and from medical records will be stored coded in an Excel data base.

Ethical Issues Data collection and handling will be coded to assure privacy of participants and will be handled by Prof. Ariel Miller and his authorized staff only. All the keys to the codes will be locked. Participants' follow-up and visits to the clinic will continue as usual. Patients' treatment will not be influenced by the study.

Intervention to promote adherence to therapy will be managed by a M.Sc. health therapist. Ethical issues of the profession will be strictly kept.

Data Management Data collected through participants and physician filled forms and from medical records will be stored coded in a data base. The database is password protected. Prof Ariel Miller and his authorized staffs are responsible for its update and data verification.

Data Analysis Data analysis will be performed using the SPSS statistical package version 22.0 (SPSS Inc., Chicago, Illinois, USA). Comparisons of continuous characteristics of adherent and non-adherent patients will be performed by Student's t-test or Mann-Whitney test, according to data distribution. Categorical variables will compared using Chi square test or Fisher's exact test for small sample.

To examine initiation and persistence of adherence to medication among patients, McNemar test or Paired T test or Wilcoxon signed ranks test will be applied as appropriate.

Multivariable Logistic regression model will be used to examine the association between illness perception and medication perception to adherence, controlling for background variables such as depression, anxiety, time since diagnosis and medical condition. Odd Ratio and 95 % confidence intervals will be calculated from the model.

The relationship between the variables in MyMS_PASS and the rates of adherence will be assessed by multiple logistic regression.

Multivariable Logistic regression model will be used to assess the influence of interventions on adherence, controlling for other parameters.

The association between the intervention and other continuous study parameters such as motivation, goals, habit formation, and quality of life will be tested with T-test or Mann-Whitney test.

Repeated measures tests will be employed to examine the effect of intervention on illness and medication perception over time.

All p values will be two-sided, and statistical significance is defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* MS patients according to Poser diagnosis
* treated or planned to be treated with Disease Modifying Therapies
* age 18 to 70
* signed informed consent
* both male and female

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-08; Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to therapy by assessment of remaining pills/medication claims electronic records | 24 months
  For oral therapy: Adherence to therapy as indicated by the number of pills remaining in the pills empty packages
Adherence to therapy according to ProMas | 24 months
  Improvement in therapy adherence as measured by Probabilistic Medication Adherence Scale (ProMas). Adherence categories are low (sum score 0-4), medium low (sum score 5-9), medium-high (sum score 10-14) and high (sum score 15-18)
Adherence to therapy according to MS-TAQ | 24 months
  Improvement in therapy adherence as measured by Multiple Sclerosis Treatment Adherence Questionnaire (MSTEQ). The items from MS-TAQ used in this analysis tapped whether the participant did not take a prescribed dose in the last four weeks and the reported number of these doses. In cases of reported non-adherence, the percentage was calculated per regiment.

SECONDARY OUTCOMES:
Improvement in quality of life | 24 months
  Improvement in quality of life as measured by the World Health Organization Quality of Life-Bref instrument (WHOQOL-Bref)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Miller, MD, PhD, Principal Investigator — Technion, Israel Institute of Technology, and Carmel Medical Center
Locations (1):
- MS Clinic, Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Neter E, Glass-Marmor L, Wolkowitz A, Lavi I, Miller A. Beliefs about medication as predictors of medication adherence in a prospective cohort study among persons with multiple sclerosis. BMC Neurol. 2021 Mar 25;21(1):136. doi: 10.1186/s12883-021-02149-0. PMID 33761887